CLINICAL TRIAL: NCT03571165
Title: Feasibility Study of an On-Line Intervention "My Tools 4 Care - In Care" for Family Caregivers of Residential-Living Older Persons With Dementia
Brief Title: Feasibility Study of "My Tools 4 Care-In Care" for Family Caregivers of Residential-Living Older Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Frailty Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00065220
Record Dates: First submitted 2018-06-17; First posted 2018-06-27 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2020-03

CONDITIONS: Dementia; Family
Keywords: carers; quality of life; dementia; web-based intervention
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention group received information on accessing My Tools 4 Care - In Care for 2 months.
  Interventions: Behavioral: My Tools 4 Care - In Care

INTERVENTIONS:
Behavioral: My Tools 4 Care - In Care — Self-administered web-based transition toolkit (My tools 4 Care - In Care) contains interactive activities and resources to help carers through transitions.

SUMMARY:
Following institutionalization of a relative with Alzheimer's disease and related dementia (ADRD), family carers continue to provide care and must learn to negotiate with staff, and navigate the system, all of which can affect their mental health. A web-based intervention, My Tools 4 Care - In Care (MT4C-In Care) will be developed to aid carers through the transitions experienced when their frail older relative/friend with ADRD resides a in Long-Term Care Facility (LTC).

A mixed method pre-post-test longitudinal feasibility study will be used to evaluate MT4C-In Care for feasibility, acceptability, ease of use, and satisfaction. In addition, the investigators expect that MT4C-In Care will improve carers hope, general self-efficacy, quality of life, and reduce their feelings of loss and grief. Following baseline data collection 40 carers of persons with ADRD will be given access to MT4C-In Care over a 2 month period. Measures will be collected at baseline, 1, and 2 months.

DETAILED DESCRIPTION:
Background: Those who are admitted to long term care facilities (LTC) often have complex health needs making them frail and vulnerable. In addition, most have dementia. Families (broadly defined to include friends) continue to provide care after their relative is admitted to LTC with the added dimensions of negotiating with staff in the provision of care and learning to navigate the system. Family caregivers of persons with dementia experience negative physical and psychological well-being as a result of caregiving and their mental health may actually worsen after the institutionalization of a family member. The research team developed and is currently testing a web-based intervention My tools 4 Care (MT4C) for carers of persons with dementia and multiple chronic conditions in the community. MT4C is an interactive toolkit intended to help caregivers with their transitions. The research team was approached by family caregivers of persons with dementia in LTC to develop a toolkit tailored to their needs. The investigators expect that this new toolkit My Tools 4 Care-In Care (MT4C - In Care) will help users through significant changes and improve caregiver outcomes.

Research Questions: 1) What revisions should be made to My Tools 4 Care to tailor it to the needs of caregivers of older frail persons with dementia residing in LTC?, 2) What are the family caregivers' perceptions of the acceptability, feasibility, ease of use, and satisfaction with the toolkit? 3) How do study participants describe their hope, general self-efficacy, loss and grief and quality of life over time while participating in the study?, and 4) What is the use and cost of health services by the study participants?

Sample: Participant recruitment will take place from January 2017 to February 2017, using several strategies. Participants from another study who consented to be contacted for future relevant studies and who had a family member with ADRD residing in LTC will be contacted. Other forms of recruitment will include newspaper ads in two cities in Alberta, Canada and the Alzheimer Society of Alberta & NWT e-newsletter along with dissemination of study pamphlets to family carers attending the organization's events.

Eligible participants will be contacted by trained Research Assistants who will explain the study and obtain verbal informed consent over the telephone to participate in the study.

Design: The study will involve 3 phases. Phase 1 will consist of focus group interviews with 6-8 family carers of persons with Alzheimer's disease and related dementias (ADRD) residing in LTC. These carers will be asked to review MT4C and answer open-ended questions to provide recommendations for change. During phase 2 MT4C-In Care will be developed based on information gathered during phase1 and input from a community advisory committee. In partnership with information technology web-developers (ATMIST), the new toolkit will be available in an online format. Phase 3 will use a mixed method pre-post-test longitudinal feasibility study. Forty carers of persons with ADRD will be given access to MT4C-In Care, following informed consent and baseline measures. Participants will be instructed to use MT4C-In Care at their convenience over a 2-month period. Information on participants use of MT4C-In Care will be collected with a checklist at 1 and 2 months. Outcome measures of hope, general self-efficacy, loss and grief, and quality of life will be collected at baseline, 1 month, and 2 months. As well, participants will be asked to complete a questionnaire at baseline and 2 months regarding their use of health and social services. Finally, at 2 months participants will complete a qualitative interview regarding the ease of use, feasibility, acceptability, and satisfaction with the toolkit and recommendations for revisions to the toolkit. All data collection will take place over the telephone and will be audio-recorded.

ELIGIBILITY:
Inclusion Criteria:

1. family/friend carer of a person with ADRD, 65 years of age or older, residing in a 24-hour care facility
2. 18 years of age or older
3. English speaking
4. access to the internet and an email account.

Exclusion Criteria:

1. family/friend of a person under the age of 65, who does not have ADRD, or who is not residing in a 24-hour care facility;
2. no internet access or email account.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the 12-item Short-Form Health Survey (SF-12v2) - Mental Component Summary Score at one and two months | baseline, 1 month, and 2 months
  The SF-12v2 is a measure of health related quality of life and provides 2 scores 1) Mental Component Summary Score (MCS) and 2) Physical Component Summary Score (PCS). MCS scores range from 0 to 100, higher scores indicate better mental health related quality of life.

SECONDARY OUTCOMES:
Change from baseline in the 12-item Short-Form Health Survey (SF-12v2) - Physical Component Summary Score at one and two months | baseline, 1 month, and 2 months
  The SF-12v2 is a measure of health related quality of life and provides 2 scores 1) Mental Component Summary Score (MCS) and 2) Physical Component Summary Score (PCS). PCS scores range from 0 to 100, higher scores indicate better physical health related quality of life.
Change from baseline in the Herth Hope Index Score (HHI) at one and two months | baseline, 1 month, 2 months
  The HHI is a 12-item Likert-type scale used to measure hope. Items are scored from 1 "strongly disagree" to 4 "strongly agree", total scores range from 12 to 48 with a higher scores indicating greater hope. The items in the scale can be further divided into three factors of hope a) temporality and future, b) positive readiness and expectancy, and c) interconnectedness. Factor scores range from 4 to 16.
Change from baseline in the General Self-Efficacy Scale (GSES) at one and 2 months | baseline, 1 month, 2 months
  The GSES is a 10 item 4-point scale. The scale assesses a person's perceived self-efficacy-their belief that they can complete novel or difficult tasks or cope with diversity. Total scores range from 10 to 40 with higher scores indicating a greater level of self-efficacy.
Change from baseline in the Non Death Revised Grief Experience Inventory (NDRGEI) at one and two months | baseline, 1 month, 2 months
  The NDRGEI is a 22 item scale scored on a 6-point Likert scale from slightly disagree to strongly agree. The scale measures the grief experiences of persons anticipating a loss through four domains a) existential concerns (scores range 6-36), b) depression (scores range from 6-36), c) tension and guilt (scores range from 3-18), and d) physical distress (scores range from 7-42). The scale also offers a total grief score by calculating the sum of the four domains. The range for the total score is 22-132; higher scores indicate lower grief.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy D Duggleby, PhD, Principal Investigator — University of Alberta
Locations (1):
- University Of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duggleby W, Jovel Ruiz K, Ploeg J, McAiney C, Peacock S, Nekolaichuk C, Holroyd-Leduc J, Ghosh S, Brazil K, Swindle J, Forbes D, Woodhead Lyons S, Parmar J, Kaasalainen S, Cottrell L, Paragg J. Mixed-methods single-arm repeated measures study evaluating the feasibility of a web-based intervention to support family carers of persons with dementia in long-term care facilities. Pilot Feasibility Stud. 2018 Oct 31;4:165. doi: 10.1186/s40814-018-0356-7. eCollection 2018. PMID 30410783